CLINICAL TRIAL: NCT05340881
Title: Systematic Light Exposure Intervention for Fatigue and Cognitive Efficiency in Pediatric Brain Tumor Survivors
Brief Title: Systematic Light Exposure in Pediatric Brain Tumor Survivors
Acronym: SLEPBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); St. Jude Children's Research Hospital (Other)
Responsible Party: Principal Investigator, Kimberly Raghubar, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H-50648; R21NR019892 (NIH)
Record Dates: First submitted 2022-03-23; First posted 2022-04-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Brain Tumor
Keywords: Pediatric Oncology; Fatigue; Cognitive Late Effects; Light Exposure; Sleep; Mood; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Fatigue | interventions — Mental Status and Dementia Tests; Neuropsychological Tests; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial design
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bright Light Exposure (Active Comparator): Participants are exposed to bright light (1,000 lux at eye level) using light glasses (Luminette Version 3) for a maximum duration of 30 minutes upon awakening each day from Monday to Friday for 6 weeks while wearing an actigraph and periodic completion of questionnaires, cognitive assessments, and lab work.
  Interventions: Behavioral: Bright Light Exposure; Other: Cognitive Assessment
- Dim Light Exposure (Placebo Comparator): Participants are exposed to exposed to dim light (equivalent intensity of <25 lux) using light glasses (Luminette) for a maximum duration of 30 minutes upon awakening each day from Monday to Friday for 6 weeks while wearing an actigraph and periodic completion of questionnaires, cognitive assessments, and lab work.
  Interventions: Behavioral: Dim Light Exposure; Other: Cognitive Assessment

INTERVENTIONS:
Behavioral: Bright Light Exposure — Research coordinator will follow-up with participant on Days 2 & 5, and weekly thereafter to assess for the presence of potential side effects. If side effects are present with bright light initiation and they do not resolve by Day 5, the intervention will be discontinued.
  Arms: Bright Light Exposure
Behavioral: Dim Light Exposure — A placebo pair of glasses that is identical in form to the bright light glasses with the exception of light intensity will be used in a manner identical to the bright light glasses.
  Other Names: Placebo
  Arms: Dim Light Exposure
Other: Cognitive Assessment — Cognitive examinations will be completed in-person and remotely via an online platform; caregivers and participants will also be asked to complete questionnaires assessing fatigue, sleep, and mood. These outcomes will be completed at baseline (prior to intervention/placebo), Week 4, Week 6 (end of intervention/placebo), and Week 8 (2-weeks post intervention/placebo).
  Other Names: Cognitive tests and questionnaires

SUMMARY:
Children and adolescents treated for a brain tumor often experience fatigue and cognitive symptoms, such as slowed information processing and inattention. These symptoms may cause difficulty carrying out daily activities at home and at school. There are few well-researched, non-pharmacological interventions aimed at improving symptoms of fatigue and by extension cognitive symptoms. Systematic bright light exposure has been shown to improve symptoms of fatigue in adult survivors of cancer and children treated for some forms of cancer. This is a pilot/feasibility study and the first known study in children treated for a brain tumor. Findings from this study will be used to help plan a larger study to examine the effectiveness of this intervention and mechanisms of action.

PRIMARY OBJECTIVE:

1. To evaluate feasibility and adherence in a study of systematic bright light exposure used to improve fatigue and cognitive efficiency in survivors of pediatric brain tumor, including rates of enrollment, adherence, and acceptability.

   SECONDARY OBJECTIVES:
2. To estimate the effect size of change in fatigue associated with bright light exposure.
3. To estimate the effect size of change in cognitive efficiency associated with bright light exposure.

DETAILED DESCRIPTION:
Participants will be randomized to take part in one of two groups:

1. The Bright Light Group will be exposed to bright light (1,000 lux at eye level) using light glasses (Luminette Version 3) for a maximum duration of 30 minutes each day from Monday to Friday for a total of 6 weeks. Duration of light exposure will be gradually increased over the first few days until the target of 30 minutes is reached on Day 5. Light duration is for 10 mins on Days 1 & 2, 20 mins on Days 3 & 4, and finally, 30 mins on Day 5.
2. The Dim Light Group will be exposed to dim light (equivalent intensity of <25 lux) for a maximum duration of 30 minutes. Dim light will be given in the same manner and frequency as described for the Bright Light group.

Participants will undergo the same evaluations and monitoring throughout the intervention and post-intervention follow-up. All participants will receive a pair of light glasses, with a phone app to track usage, and be fitted with an actigraph following consent to participate. Assessments will be completed at baseline (prior to intervention), with additional assessments at Week 4 (of intervention), Week 6 (end of intervention), and 2-weeks post-intervention (Week 8). Participants and their caregivers will complete questionnaires assessing fatigue, sleep, and mood. Psychological testing to measure attention, working memory, executive control, and processing speed will be completed using a computerized, online battery at each time point and in person at baseline and end of intervention. Caregivers will also be asked to complete a questionnaire about the family's general characteristics and medical history.

At baseline and end of intervention (Week 6), saliva will be collected. For each day of the intervention, participants will share their usage data and complete a daily sleep diary that includes time spent in bed, sleep/wake times, estimated amount of natural sunlight exposure, and medication use. A research coordinator will contact families on Days 2 and 5 and weekly thereafter for the duration of the intervention to identify possible light-related side effects and to check on compliance with light exposure (both frequency and duration). A remote app will be installed on the participant's or caregiver's cell phone to share light usage, which is tracked automatically once the device is turned on. At end of intervention (Week 6), participants and their caregivers will be asked to complete a short acceptability questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and treated for a brain tumor at Texas Children's Hospital
* Treated with either surgery only or surgery and proton beam radiation therapy
* Treated for tumors other than high-grade gliomas, brain stem gliomas, or atypical teratoid rhabdoid tumors given associated reduced survival rates
* Currently or previously enrolled in longitudinal studies of neurocognitive outcomes in survivors of pediatric brain tumor (Lisa Kahalley, PI; H-29026, H-35681, H-40804, H-40961, H-49380, H-26785, H-41705
* Ages 10-18 years
* At least 1 year post-diagnosis
* Endorsed mild to moderate symptoms of fatigue on the PROMIS
* Approval from Long-Term Survivorship provider
* Adequate vision for computerized tasks
* English-speaking
* Intelligence Quotient (IQ) above 70

Exclusion Criteria:

* Diagnosis and/or treatment for secondary malignancy in the past 12 months
* Current or previous (within 12 months) suicidal ideation or severe depression requiring immediate intervention
* Presence of photophobia or other eye diseases, seizures, and/or migraines
* Use of photosensitizing medications
* Current or previous use of light therapy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent of approached participants who consent to study participation | Once, prior to enrollment
  The rates of study participation and related 90% Blyth-Still-Casella intervals, as well as their regular 90% confidence interval, will be estimated. Test of one proportion will be performed against an estimated rate of 70%. The rate will be evaluated for the group as a whole as well as separately for the bright light intervention and placebo-control groups.
Percent of sessions completed during all 6 weeks of bright or dim light exposure | At completion of bright or dim light exposure (Week 6)
  The rates of light intervention adherence and related 90% Blyth-Still-Casella intervals, as well as their regular 90% confidence interval, will be estimated. Test of one proportion will be performed against an estimated rate of 77% of sessions completed on average. The rate will be evaluated for the group as a whole as well as separately for the bright light intervention and placebo-control groups.
Percent of participants rating the intervention as acceptable by indicating that they would recommend this intervention to other survivors. | Once, at completion of intervention (Week 6)
  The rates of completion of cognitive assessments and related 90% Blyth-Still-Casella intervals, as well as their regular 90% confidence interval, will be estimated. Test of one proportion will be performed against an estimated rate of 75%. The rate will be evaluated for the group as a whole as well as separately for the bright light intervention and placebo-control groups.

SECONDARY OUTCOMES:
Change in fatigue outcome | Baseline (prior to start of intervention) compared to Week 4 (common length of intervention in adult literature)
  For the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale, the raw score is converted to a standardized T-score (range 34-85) with a mean of 50 and standard deviation of 10, where a higher score represents greater severity of symptoms. The effect size (Cohen's d- the standardized difference between two means) of bright light exposure on fatigue will be estimated by comparing performance at baseline to that at Week 4 (comparison point in adult literature), using the paired difference divided by its estimated standard deviation. In addition, given potential for missing data, a mixed-effect model will be fit to investigate change in outcome from baseline to Week 4.
Change in fatigue outcome | Baseline (prior to start of intervention) compared to Week 6 (end of intervention)
  For the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale, the raw score is converted to a standardized T-score (range 34-85) with a mean of 50 and standard deviation of 10, where a higher score represents greater severity of symptoms. The effect size (Cohen's d- the standardized difference between two means) of bright light exposure on fatigue will be estimated by comparing performance at baseline to that at Week 6 (end of systematic light exposure), using the paired difference divided by its estimated standard deviation. In addition, given potential for missing data, a mixed-effect model will be fit to investigate change in outcome from baseline to Week 6.
Change in neurobehavioral outcome | Baseline (prior to start of intervention) compared to Week 4 (common length of intervention in adult literature)
  Attention serves as the primary neurobehavioral endpoint, and it is measured by Omissions T-score (M = 50, SD = 10) from the Conners Continuous Performance Test, Third Edition (CPT-3), where higher scores indicate worse performance (<45 is low and 70+ is very elevated). The effect size (Cohen's d- the standardized difference between two means) of bright light exposure on attention will be estimated by comparing performance at baseline to that at Week 4 (comparison point in adult literature), using the paired difference divided by its estimated standard deviation. In addition, given potential for missing data, a mixed-effect model will be fit to investigate change in outcome from baseline to Week 4.
Change in neurobehavioral outcome | Baseline (prior to start of intervention) compared to Week 6 (end of intervention)
  Attention serves as the primary neurobehavioral endpoint, and it is measured by Omissions T-score (M = 50, SD = 10) from the Conners Continuous Performance Test, Third Edition (CPT-3), where higher scores indicate worse performance (<45 is low and 70+ is very elevated). The effect size (Cohen's d- the standardized difference between two means) of bright light exposure on attention will be estimated by comparing performance at baseline to that at Week 6 (comparison point in adult literature), using the paired difference divided by its estimated standard deviation. In addition, given potential for missing data, a mixed-effect model will be fit to investigate change in outcome from baseline to Week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly P Raghubar, PhD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital; Heather M Conklin, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified data for all IPD that underlie results in a publication upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication.
Access Criteria: Upon request to PI